CLINICAL TRIAL: NCT03221686
Title: The Effect of a Pre- and Postoperative Oral Supplement of Arginine, Zinc and Vitamin C on Collagen Synthesis in Surgical Inguinal Hernia Patients: A Randomized Controlled Trial
Brief Title: Effects of Oral Supplementation of Arginine, Zinc and Vitamin C on Collagen Synthesis in Inguinal Hernia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lars Nannestad Jorgensen (Other)
Responsible Party: Sponsor-Investigator, Lars Nannestad Jorgensen, Professor, MD, DrMedSci, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H-15017272
Record Dates: First submitted 2017-03-30; First posted 2017-07-18 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2017-07

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Total daily protein intake: 1.5 g protein/kg body weight
  Interventions: Dietary Supplement: Control
- Intervention (Active Comparator): 55 mg zinc/day, 1251 mg vitamin C/day, and 15 g arginine/day. Total daily protein intake: 1.5 g protein/kg body weight
  Interventions: Dietary Supplement: Intervention

INTERVENTIONS:
Dietary Supplement: Intervention — The patients in the intervention group are given 55 mg zinc, 1251 mg vitamin C, and 15 g arginine once daily 14 days pre-operatively and post-operatively together with a high quality protein supplement.
  Arms: Intervention
Dietary Supplement: Control — High quality protein supplement 14 days pre-operatively and post-operatively.
  Arms: Control

SUMMARY:
Collagen synthesis is depressed systemically in the immediate postoperative period. Arginine, zinc and vitamin C impact collagen synthesis.

The aim of this study is to investigate the effect of a pre and postoperative oral supplement consisting of arginine, zinc and vitamin C on collagen synthesis in patients undergoing inguinal hernia repair.

DETAILED DESCRIPTION:
The trial investigates the effect of a pre and postoperative oral supplement consisting of arginine, zinc and vitamin C on collagen type I synthesis in patients undergoing inguinal hernia repair.

The patients in the intervention group are given 55 mg zinc, 1251 mg vitamin C, and 15 g arginine once daily 14 days pre-operatively and post-operatively. Both groups receive high quality protein (1.5 g protein/kg body weight) daily during the same period. Hernia repair is done using the Lichtenstein technique. Drainage tubes are placed in the wound during the surgery. Epidermal wounds (10 mm) are made via the suction blister method on the ventral forearm of the patients on the day of surgery. Blood samples are drawn at day -14, day 0, day 1 and day 2. The surgical drain is emptied and fluid collected at day 1 and day 2.The healing of the suction blisters is assessed by clinical criteria until healing.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* Patients undergoing hernia repair using the Lichtenstein technique
* Written informed consent

Exclusion Criteria:

* Former surgery in the same area within 5 years
* Dementia
* Dysregulated diabetes
* Systemic corticosteroid treatment
* Liver disease
* Kidney disease
* Cancer within 5 years
* Need of interpreter

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-02-20 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-12-10 (Actual)

PRIMARY OUTCOMES:
Changes in CICP levels in serum. CICP is the biomarker of type I collagen synthesis (carboxy-terminal propeptide of type I procollagen) | Day 2
  CICP is measured by enzyme-linked immunosorbent assay

SECONDARY OUTCOMES:
Changes in CICP levels in wound fluid collected from surgical drain. CICP is the biomarker of type I collagen synthesis (carboxy-terminal propeptide of type I procollagen). | Day 1 and day 2
  CICP is measured by enzyme-linked immunosorbent assay
Changes in CICP levels in wound fluid collected from suction blisters. CICP is the biomarker of type I collagen synthesis (carboxy-terminal propeptide of type I procollagen). | Day 0
  CICP is measured by enzyme-linked immunosorbent assay
Changes in Zinc levels in serum | Day -14, day 0, day 1 and day 2
  Zinc is measured by direct spectrophotometry
Changes in Zinc levels in wound fluid collected from surgical drain | Day 1 and day 2
  Zinc is measured by direct spectrophotometry
Changes in Zinc levels in wound fluid collected from suction blisters | Day 0
  Zinc is measured by direct spectrophotometry
Changes in Arginine levels in serum | Day -14, day 0, day 1 and day 2
  Arginine is measure by ultra-performance liquid chromatography and mass spectrometry
Healing of suction blisters | Day 3 to Suction Blister healing
  Clinical assessment
Compliance | Day -14 to Suction Blister healing
  Count of remaining supplement

CONTACTS AND LOCATIONS:
Overall Officials: Lars N Joergensen, Principal Investigator — K. Forskning, BIspebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Copenhagen NV, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kjaer M, Frederiksen AKS, Nissen NI, Willumsen N, van Hall G, Jorgensen LN, Andersen JR, Agren MS. Multinutrient Supplementation Increases Collagen Synthesis during Early Wound Repair in a Randomized Controlled Trial in Patients with Inguinal Hernia. J Nutr. 2020 Apr 1;150(4):792-799. doi: 10.1093/jn/nxz324. PMID 31897483